CLINICAL TRIAL: NCT06234254
Title: Reducing Adult Inpatients Anxiety With Virtual Reality Meditation: A Prospective, Randomized Study
Brief Title: Reducing Adult Inpatients Anxiety With Virtual Reality Meditation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 73841
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Virtual Reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants will be immersed in a virtual environment. Calming scenery will be shown via the headset for 20-30 minutes
  Interventions: Behavioral: Virtual Reality headset with calming scenery
- Control (No Intervention): No intervention (i.e. virtual reality headset) will be applied to the participant.

INTERVENTIONS:
Behavioral: Virtual Reality headset with calming scenery — Participants will be immersed in a virtual environment. Calming scenery will be shown via the headset for 20-30 minutes
  Arms: Virtual Reality

SUMMARY:
The purpose of the study is to evaluate if non-invasive, distracting devices (virtual reality) can decrease anxiety and improve affect and satisfaction in adult, hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* between age 18-99
* hospitalized at Stanford Health Care
* english-speaking

Exclusion Criteria:

* significant cognitive impairment or inability to consent
* current nausea
* visual problems or currently using corrective glasses that are incompatible with the virtual reality headset
* a history of severe motion sickness
* a history of seizures cause by flashing light
* clinically unstable or require immediate/urgent intervention

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Before and Immediate after intervention
  Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Caruso, Study Director — Stanford University
Locations (1):
- Stanford Health Care (SHC), Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No